CLINICAL TRIAL: NCT07397468
Title: Double-blind, Placebo-controlled, Randomized, Safety and Efficacy Study of JUV-161 Administered to Healthy Volunteers Undergoing Unilateral Lower Limb Immobilization (ULLI)
Brief Title: To studyJUV-161 Administered to Healthy Volunteers Undergoing Unilateral Lower Limb Immobilization (ULLI)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Juvena Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JUV161-201
Record Dates: First submitted 2026-01-27; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: double-blind, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: quadruple
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- JUV-161 5mg/kg (Experimental): Participants will receive JUV-161 5 mg/kg administered subcutaneously Each subject will receive 7 doses in total over 6 weeks.
  Interventions: Drug: JUV-161
- JUV-161 10 mg/kg (Experimental): Participants will receive JUV-161 at a dose of 10 mg/kg administered subcutaneously, contingent upon Safety Committee approval for dose escalation. Each participant will receive a total of 7 doses over a 6-week dosing period.
  Interventions: Drug: JUV-161
- Placebo (Placebo Comparator): Participants will receive matched placebo administered subcutaneously. Each participant will receive a total of 7 doses over a 6-week dosing period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JUV-161 — JUV-161 administered subcutaneously at protocol-specified dose levels.
  Arms: JUV-161 10 mg/kg; JUV-161 5mg/kg
Drug: Placebo — Matched placebo administered subcutaneously
  Other Names: Matched Placebo
  Arms: Placebo

SUMMARY:
This is a double-blind, placebo-controlled, randomized study of 96 days total duration to assess the effect of JUV-161 on muscle disuse atrophy. This will be a multicenter study in New Zealand and will include up to 40 healthy volunteers aged between 40 to 65 years of age. Following the screening period, subjects will be randomized to receive either weekly subcutaneous (SC) injections of one of two doses of JUV-161 or matching placebo for a period of approximately 6 weeks.

DETAILED DESCRIPTION:
JUV-161 is being developed for the treatment of muscle atrophy or sarcopenia and myotonic dystrophy. This study is investigating the safety and efficacy of JUV-161 administered in healthy participants who are undergoing unilateral lower limb immobilization (ULLI). Muscle atrophy is a general term to describe loss of muscle mass, whereas sarcopenia is a more specific term used to describe age-related loss of muscle. Muscle atrophy can be associated with a multitude of causes ranging from poor nutrition to neurological diseases, myopathies or disuse.

JUV-161 is an agonist designed to activate key signaling pathways in skeletal muscle, promoting muscle growth, maintenance, and strength, and may help prevent muscle atrophy during periods of immobilization. ULLI or unilateral lower limb suspension (ULLS) is often the consequence of common injuries such as falls, fractures or joint injuries. Because it isolates a specific group of muscles, it is also a frequently used model to study muscle disuse atrophy. In fact, ULLI/S using a brace or cast is the most frequent model used to study disuse atrophy.

This is a double-blind, placebo-controlled, randomized multicenter study of 96 days total duration. The purpose is to assess the effect of JUV-161 on muscle disuse atrophy. The study will include up to 40 healthy volunteers aged between 40 and 65 years of age (inclusive). Following the screening period, subjects will be randomized 1:1 to receive either weekly subcutaneous (SC) injections ofJUV-161 or a matching placebo for a period of approximately 6 weeks (total of 7 doses).

The study will be conducted in three phases:

* Immobilization to induce disuse muscle atrophy. Subjects will have one leg immobilized using a brace and boot to prevent weight bearing. (Crutches will be provided). The leg will be immobilized for 14 days, then the brace/boot will be removed.
* Recovery (mobilization) After the brace/boot is removed, subjects will undergo a 4-week period of mobilization to help restore muscle mass and strength lost in the immobilized leg
* Resistance exercise training (RET) After 4 weeks of mobilization, subjects will undergo a further 3 weeks of personalized (RET) to fully restore muscle mass and strength in the immobilized leg. Participants and researchers will be blinded to the study allocation. Every person in the study will have their dominant leg fitted with a brace, which they will wear for 15 days. They will then receive 5mg/kg of the JUV-161 (or matching placebo) once a week for 6 weeks (7 doses total). This will be given as a subcutaneous (SC) injection in the abdomen or thigh. The study design includes an option for a single escalation of the JUV-161 dose based on SRC review of blinded aggregate safety data after 18 participants in the initial dose group have completed the first 14 days of treatment with study drug.

If dose escalation is supported, no further participants will be enrolled in the initial dosing group, and 18 subjects will be enrolled in the higher dose group. If dose escalation is not supported by safety data, enrollment of further participants will continue in the initial dosing group until a total of 36 subjects have been enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Males or post-menopausal females aged ≥40 years of age and ≤65 years of age at time of informed consent. Post-menopausal is defined as no menses for at least 12 months without an alternative medical cause and a Screening follicle stimulating hormone (FSH) level >40 U/L.
2. Willing and able to give informed consent and comply with the requirements of the protocol, including muscle biopsy.
3. Are healthy in the opinion of the Investigator, based on physical examination, medical history, clinical laboratory tests, vital signs, and resting electrocardiogram.
4. BMI ≤ 30 kg/m2
5. Ambulatory (N.B.: The study may not suitable for subjects who need to drive or have dependents who require them to be fully mobile or difficult access to home or work.)

Exclusion Criteria:

1. Any anabolic steroid use or any condition that might affect muscle mass or strength
2. Participation in resistance or strength training at a frequency >1 time/week within 30-days prior to screening
3. Weight-loss diet within 30-days prior to screening or actively pursuing weight loss, or intending to actively pursue weight loss diet or activities during the study.
4. Use of dietary supplements e.g. protein supplements, amino-acid supplements within 30 days prior to Screening: use of protein supplements within 4 weeks prior to randomization; use of omega-3 supplements within 3 months prior to Screening.
5. History of alcohol misuse (males: ≥14 standard drinks/week, females ≥7 standard drinks/week) or drug misuse (current or past-12-month substance use disorder per DSM-5 and/or ICD criteria).
6. Have an active malignancy or have a history of malignancy within 5 years prior to Screening. (Subjects with prior basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that were successfully treated may be included.)
7. Have any of the following known active infections:

   1. Infection requiring systemic antiviral or antimicrobial therapy that will not be completed within 30 days prior to screening
   2. Known history of, or positive Screening serology test result for, any of Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV).
8. Have any clinical history or other active medical condition, psychiatric disorder or clinically significant laboratory abnormality, vital sign, ECG abnormality or other finding that, in the investigator's opinion, is likely to increase the risk of study participation, confound study results, interfere with study conduct, or otherwise risk non-compliance with study requirements.
9. Implanted electronic device e.g. pace-maker, ICD, nerve stimulator, infusion pump.
10. Have any of the following:

    1. History of diabetes, thyroid disease, liver disease, coronary artery disease, peripheral vascular disease or risk factors for peripheral vascular disease (e.g., uncontrolled hypertension, obesity, diabetes, hypercholesterolemia > 6.5 mmol/L (250 mg/dl), claudication or evidence of venous or arterial insufficiency upon palpitation of femoral, popliteal and pedal arteries)
    2. History of bleeding disorder or excessive bleeding
    3. At risk for, or previous history of deep vein thrombosis (DVT) (including family history)
    4. History of pulmonary emboli
    5. History of myeloproliferative disease including polycythemia vera (Hb >16.5 g/dL for males or >16.0 g/dL for females and/or hematocrit >49% for males or >48% for females) or thrombocytosis (platelet count >400 x109/L)
    6. History of connective tissue diseases (positive lupus anticoagulant), hyperhomocysteinemia, deficiencies of factor V Leiden, proteins S and C, and antithrombin III
    7. Impaired renal function (estimated glomerular filtration rate [eGFR] <60ml/min/1.73m2, using the CKD-EPI (2021) equation)
    8. Platelet count < 125 X 109/L
    9. Use of anticoagulants or INR > ULN
    10. Electrocardiogram (ECG) showing QTcF > 470 msec female or > 450 msec male
11. Have received treatment with any prescription medication or treatment with any non-prescription medication within 14 days prior to screening (exception: acetaminophen up to 2 g per day prior to dosing is permitted) The use of statins, steroids or non-steroidal anti-inflammatory agents is specifically prohibited.
12. Any vaccination (therapeutic or prophylactic) within 30 days prior to screening and/or plans to receive any vaccination during the course of the study.
13. Prior exposure to JUV-161 or have known allergies to any components of the JUV-161 formulation.
14. History of immune reaction to any biologic therapy.
15. Donation or loss of greater than 1 unit (450 mL) of blood or donation of plasma through plasmapheresis within 30 days prior to screening.
16. Pregnant, breast-feeding, or is a woman of child-bearing potential (defined as fertile and following menarche until becoming post menopausal) or is not confirmed as post-menopausal at screening.
17. Use of hormone therapy e.g. estrogen within 60 days before Screening.
18. Recent (within 3 months of screening) history of surgery or significant trauma.
19. Active smoker or history of smoking/ nicotine use within the last 5 years before screening, and/or unwilling to abstain from tobacco/nicotine use during the study.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | from enrollment through to Day 96
Number of Participants who have Change in Quadriceps Muscle Mass and Volume as assessed by magnetic resonance imaging MRI. | Change from baseline (pre-treatment) to Day 15 (post-immobilization) and Day 45 (post-treatment)
Number of participants who have Change in lower limb muscle architecture as assessed by MRI. | Change from baseline (pre-treatment) to Day 15 (post-immobilization) and Day 45 (post-treatment)
  includes individual muscle volume, intramuscular fat fraction, spatial distribution of fat fraction, and quantification of short tau inversion recovery (STIR) hyperintensity,

SECONDARY OUTCOMES:
Change from baseline in pharmacodynamic biomarkers of target engagement (myostatin and follistatin) | Change from baseline (pre-treatment) to Day 15 (post-immobilization) and Day 45 (post-treatment)
  Change from baseline in serum concentrations of myostatin and follistatin, measured using validated immunoassays.
Change from baseline in myogenesis-related biomarkers (IGF-1 and human growth hormone) | Change from baseline (pre-treatment) to Day 15 (post-immobilization) and Day 45 (post-treatment)
  Change from baseline in serum concentrations of insulin-like growth factor-1 (IGF-1) and human growth hormone, measured using validated immunoassays.
Change from baseline in metabolic and inflammatory biomarkers (IL-6, TNF-α) | Change from baseline (pre-treatment) to Day 15 (post-immobilization) and Day 45 (post-treatment)
  Change from baseline in serum concentrations of interleukin-6 (IL-6) and tumor necrosis factor alpha (TNF-α), measured using validated immunoassays.

OTHER OUTCOMES:
Number of participants who have Change in Lower Limb Muscle Strength as assessed by isokinetic dynamometry (force output). | Change from baseline (pre-treatment) to Day 15 (post-immobilization) and Day 45 (post-treatment)
Number of Participants who have Change in Lower Limb Force Production as assessed by single-leg vertical jump height. | Change from baseline (pre-treatment) to Day 15 (post-immobilization) and Day 45 (post-treatment)
Number of participants who have Change in Lower Limb Muscle Fatigue as assessed by single-leg vertical jump height | hange from baseline (pre-treatment) to Day 15 (post-immobilization) and Day 45 (post-treatment)
Number of participants who have Change in Muscle Protein Synthesis Rate as measured in vastus lateralis muscle biopsy samples | Change from baseline (pre-treatment) to Day 15 (post-immobilization) and Day 45 (post-treatment)
Number of participants who have Change in lower limb muscle architecture as assessed by ultrasound | Change from baseline (pre-treatment) to Day 15 (post-immobilization) and Day 45 (post-treatment)
Number of participants who have Changes in metabolic profile via glucose and calculated insulin sensitivity | Change from baseline (pre-treatment) to Day 15 (post-immobilization) and Day 45 (post-treatment)
Maximum observed plasma concentration (Cmax) | Day 1 pre-dose and at 1, 2, 6, 12, 24, 36, 48, 72 on Days 1,15,45
Time to the maximum measured plasma concentration (Tmax): | Up to 48 days
Area under the concentration-time curve from time zero through to infinity (AUC0-∞) | Up to 48 days
Terminal elimination half-life in plasma (t1/2) | Up to 48 days
Presence and titers of anti-drug antibodies (ADAs) and identification of neutralizing antibodies (NAbs). | Up to 96 Days

IPD SHARING:
Plan to Share IPD: No